CLINICAL TRIAL: NCT01785017
Title: The Effects of a Standardized Clinical Assessment Management Plan (SCAMP) on Clinical Outcomes in Children With Critical Asthma
Brief Title: The Effects of a Standardized Management Plan on Children With Critical Asthma
Acronym: AsthmaSCAMP
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jackson Wong, MD, Boston Children's Hospital
Other Study IDs: 00006397
Record Dates: First submitted 2013-01-31; First posted 2013-02-06 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2013-02

CONDITIONS: Children; Asthma
Keywords: critical; asthma; children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chidren with critical asthma: Pre- and post-SCAMP

SUMMARY:
A Standardized Clinical Assessment Management Plan (SCAMP) has been developed and implemented at Boston Children Hospital to decrease variations in clinical practice in critical asthma therapies for children. The primary aim is to determine whether a Critical Asthma SCAMP can improve clinical outcome.

DETAILED DESCRIPTION:
A Standardized Clinical Assessment Management Plan (SCAMP) has been developed and implemented at Boston Children Hospital to decrease variations in clinical practice in critical asthma therapies for children. However the effects of the Critical Asthma SCAMP on the clinical outcomes in children with critical asthma are unknown. This study will assess the effectiveness of the SCAMP by comparing retrospective data from medical records in children with critical asthma to prospective clinical PPSQ SCAMP outcome data obtained during the QA process of the SCAMP. The primary aim is to determine whether a Critical Asthma SCAMP can improve clinical outcome. There are three specific pathways in the Critical Asthma SCAMP. The primary outcome measure is the length of intensive care length of stay (defined as time to every 2 hr intermittent albuterol nebulization) for all three pathways. The secondary aim is to validate a clinical asthma score to direct critical asthma therapies. To achieve this goal we will determine the relationships of the driver(s) of the SCAMP which includes Boston Children Hospital (BCH) Asthma Severity Score [HASS] and non-invasive measures of pCO2 to standard measures of severity of asthma (blood gases and peak flow measurements).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients 2 years and older requiring critical asthma therapies including continuous albuterol nebulization

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized children 2 years and older requiring intensive care treatment for asthma
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Time from initialization of continuous albuterol to time of final every 2 hr albuterol nebulization | The time to intermittent q2 hr albuterol nebulization from continuous albuterol during hospitalization within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jackson Wong, MD, Principal Investigator — Boston Children Hospital
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States